CLINICAL TRIAL: NCT07388563
Title: A Phase I Trial of Azacitidine and Abatacept in Relapsed or Refractory T-Cell Lymphoma
Brief Title: Azacitidine and Abatacept in Relapsed or Refractory T-Cell Lymphoma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10002363; 002363-C
Record Dates: First submitted 2026-02-04; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-28

CONDITIONS: Lymphoma, T Cell, Peripheral; T-cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Anaplastic Large Cell Lymphoma; Monomorphic Epitheliotropic Intestinal T-cell Lymphoma; Adult T-cell Leukemia/Lymphoma
Keywords: Selective Costimulation Modulators; Immunomodulators; Biological Therapy; Chemotherapy
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Lymphoma, T-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — Azacitidine; Abatacept

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Escalating/de-escalating doses of azacitidine + abatacept
  Interventions: Drug: azacitidine; Drug: abatacept
- Arm 2 (Experimental): MTD of azacitidine + abatacept if less than 12 participants are enrolled in Arm 1
  Interventions: Drug: azacitidine; Drug: abatacept

INTERVENTIONS:
Drug: azacitidine — Days 1-5 or 1-7 of every cycle (12 cycles): azacitidine subcutaneous or IV at the dose of 75 mg/m2
Drug: abatacept — Cycle 0, Days 1 and 15: abatacept IV infusions at the dose of 5 mg/kg or 10 mg/kg. Cycles 1-6, Day 1: abatacept IV infusions at the dose of 5 mg/kg or 10 mg/kg.

SUMMARY:
Background:

T-cell lymphoma is a blood cancer that affects immune system cells. People tend to survive less than 1 year if this disease does not respond to treatment (is refractory) or comes back after treatment (relapses). Azacitidine and abatacept are 2 drugs that are used to treat other diseases. Researchers want to know if these drugs, used together, can help people with T-cell lymphoma.

Objective:

To learn if azacitidine combined with abatacept can shrink tumors in people with T-cell lymphoma.

Eligibility:

People aged 18 years and older with T-cell lymphoma that either came back or did not respond to treatment.

Design:

Participants will be screened. They will have a physical exam with blood tests. They will have a test of their heart function. They will have imaging scans of their tumors. A sample of tumor tissue may be taken.

Azacitidine is injected under the skin of the thigh, abdomen, or upper arm. Abatacept is infused through a needle inserted into a vein in the arm.

Participants will receive the study drugs in 28-day cycles for up to 13 cycles. They will come to the clinic for each treatment. They will come to the clinic on day 1 and day 15 of the first cycle. After that, they will come to the clinic on the first 5 or 7 days of each cycle. Each clinic visit will take no more than 8 hours.

Imaging scans and other tests will be repeated during the study. Participants will have follow-up visits for up to 5 years after they stop taking the study drugs....

DETAILED DESCRIPTION:
Background:

* Relapsed or refractory T-cell lymphoma is typically incurable with a median survival of less than 1 year. Angioimmunoblastic T-cell lymphoma (AITL) is the most commonly defined subtype of T-cell lymphoma and has a similarly poor prognosis.
* We have developed the first AITL cell lines that maintain immunophenotypic fidelity with AITL and used these cell lines to identify novel therapies for patients with AITL.
* We found that CD28 blockade with the Food and Drug Administration (FDA)-approved rheumatologic agent abatacept, which blocks CD28 signaling, impaired the proliferation of AITL cell lines, and that injection of abatacept into patient-derived xenograft (PDX) models of AITL significantly prolonged their survival. Based on this we conclude that targeting CD28 with abatacept in AITL is a promising, novel therapeutic approach that warrants clinical testing in people with relapsed/refractory (R/R) T-cell lymphoma.
* Abatacept can be combined with the deoxyribonucleic acid (DNA) methyltransferase inhibitor azacitidine, which has been shown to be preferentially active in patients with a TET2 mutation, the most common genetic abnormality in patients with AITL. We confirmed that azacitidine indeed inhibits AITL cell lines synergistically with abatacept.

Objectives:

* Arm 1: To estimate the maximum tolerated dose (MTD) of the combination of azacitidine and abatacept in relapsed or refractory T-cell lymphoma.
* Arm 2: To estimate the complete response rate (CRR) of the combination of azacitidine and abatacept.

Eligibility:

* Participants >= 18 years with relapsed or refractory T-cell lymphoma after initial systemic treatment.
* Adequate organ and marrow function.
* Eastern Cooperative Oncology Group (ECOG) performance status <= 2.

Design:

* This is a non-randomized, open-label, single-site phase I trial evaluating the combination of azacitidine and abatacept.
* Treatment will be delivered in cycles consistent of 28 days.
* During Cycle 0 abatacept will be administered intravenously on Days 1 and 15.
* During Cycles 1-6 abatacept administered on Day 1 will be combined with subcutaneous azacitidine delivered on Days 1-5 or Days 1-7.
* After Cycle 6 participants will be evaluated and participants who have a response will get additional 6 cycles of the monotherapy with azacitidine.

ELIGIBILITY:
-INCLUSION CRITERIA

1. Participants must have a histologically or cytologically confirmed T-cell lymphoma confirmed by the Laboratory of Pathology (LP), NCI. The one of the following T-cell lymphomas are included:

   * Peripheral T-cell lymphoma not otherwise specified (PTCL, NOS)
   * Angioimmunoblastic T-cell lymphoma (AITL)
   * T-follicular helper (TFH) lymphoma
   * Anaplastic large cell lymphoma (ALCL)
   * Enteropathy-associated T-cell lymphoma (EATL)
   * Monomorphic epitheliotropic intestinal T-cell lymphoma (MEITL)
   * Adult T-cell leukemia/lymphoma (ATLL)
   * Other T-cell lymphoma (TCL)
2. Participants must have a disease that is relapsed or refractory after initial systemic treatment.
3. Participants must have evaluable disease on screening imaging or by laboratory assessment.
4. Age >= 18 years.
5. ECOG performance status <= 2.
6. Participants must have adequate organ and marrow function as defined below:

   * Absolute neutrophil count (ANC) / >= 1,000 cells/mcL OR >= 500 cells/mcL if bone marrow involvement with lymphoma
   * Platelets / >= 50,000 cells/mcL OR >= 25,000 cells/mcL if bone marrow involvement with lymphoma
   * Hemoglobin / >= 8 g/dL (transfusions permitted)
   * Renal function / Serum creatinine <= 2 mg/dL OR Glomerular filtration rate (GFR) >= 40 mL/min/1.73 m^2 as estimated by the Modification of Diet in Renal Disease (MDRD).

   Note: there is no limit if involved by lymphoma.

   If not on target, a 24-hour urine creatinine clearance can be used to directly measure creatinine clearance.
   * Total bilirubin / <= 1.5 x upper limit of normal (ULN)
   * Aspartate Aminotransferase (AST) / <= 3.0 x ULN
   * Alanine Aminotransferase (ALT) / <= 3.0 x ULN
   * Prothrombin time (PT) / <1.5 x ULN
   * Activated partial thromboplastin time (aPTT) / <1.5 x ULN; < 5.0 x ULN if the aPTT is prolonged because of a positive Lupus Anticoagulant

   International normalized ratio (INR) / <1.5 x ULN
7. Participants, seropositive for human immunodeficiency virus (HIV), must have an undetectable HIV viral load.
8. Participants, seropositive for hepatitis C virus (HCV) infection, must have been treated and have an undetectable HCV viral load.
9. Participants who are hepatitis B core antibody (HBcAb) positive must have a hepatitis B virus (HBV) viral load result <100 IU/mL. Note: participants who are hepatitis B surface antigen (HBsAg) positive are excluded.
10. Participants with detectable Epstein-Barr virus (EBV) or Cytomegalovirus (CMV) by polymerase chain reaction will be eligible provided they do not have end organ dysfunction from EBV or CMV infection.
11. Participants with pulmonary disease such as chronic obstructive pulmonary disease and non-infectious liver disease who otherwise meet the requirements.
12. Women of child-bearing potential (WOCBP) must agree to use effective methods of contraception (barrier, hormonal, surgical sterilization, abstinence) during the study treatment and for 6 months after the completion of the study treatment. Note: WOCBP is defined as any woman who has experienced menarche and who has not undergone successful surgical sterilization or who is not postmenopausal.

    Men able to father a child must agree to use an effective method of contraception (barrier, surgical sterilization, abstinence) during the study treatment and for 3 months after the completion of the study treatment. These men must not freeze or donate sperm within the same period.
13. Nursing participants must be willing to discontinue nursing from study treatment initiation through six (6) months after the last dose of the study drug(s).
14. Ability of the participant to understand and the willingness to sign a written informed consent document.

Exclusion Criteria

1. Any second malignancy that requires current active systemic therapy.
2. Latent tuberculosis (TB) infection.
3. Active systemic bacterial, viral, fungal, mycobacterial, parasitic, or other infection requiring anti-infective treatment within 1 day prior to the study treatment initiation.
4. Anti-cancer therapy within 2 weeks prior to the study treatment initiation. Note: systemic steroids are allowed if <= 100 mg/per day of prednisone (or equivalent) and were used for <= 7 days during 2 weeks before the study treatment initiation.
5. Any investigational therapy within 2 weeks prior to the study treatment initiation.
6. Known allergy or hypersensitivity to any of the study drugs.
7. Pregnancy confirmed with beta-human chorionic gonadotropin (beta-HCG) serum or urine pregnancy test in WOCBP at screening.
8. Active central nervous system involvement with lymphoma. Previously treated central nervous system involvement with lymphoma will be allowed if >3 months since end of treatment.
9. Uncontrolled intercurrent illness, factors, evaluated by medical history, electrocardiogram (EKG), and physical exam that would potentially increase in risk of participant.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Arm 2: To estimate the CRR of the combination of azacitidine and abatacept. | Day 1 of Cycles 1, 4, 7, 10, EOT/PD visit, every 3 months for years 1-2, every 6 months for years 3-4, once a year for year 5.
  Complete response rate (CRR) will be evaluated in Arm 2 in participants treated at MTD. CRR will be estimated along with a 95% confidence interval (CI).
Arm 1: To estimate the MTD of the combination of azacitidine and abatacept in relapsed or refractory T-cell lymphoma. | 56 days (cycles 0-1)
  MTD will be determined based on the DLT profile during the DLT window in Arm 1 56 days (cycles 0-1).

SECONDARY OUTCOMES:
To determine the ORR defined as CR + PR to the combination of azacitidine and abatacept | Day 1 of every cycle then at the EOT/PD visit, every 3 months for years 1-2, every 6 months for years 3-4, then once a year until progression, initiation of another line of therapy, or 5 years since treatment initiation.
  ORR will be estimated along with a 95% CI. Every report of response rates will contain all participants included in the study.
To determine the safety profile of a combination of azacitidine and abatacept in relapsed or refractory T-cell lymphoma | Day 1 through 30 days after the last study intervention was administered or before the initiation of a new anti-cancer treatment, whichever comes first.
  The number and frequency of adverse events for participants as assessed per CTCAE version 6. Safety will be analyzed by reporting the number of patients experiencing toxicity, classified by type and maximum grade to the experimental regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Max J Gordon, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the NIH Data Management and Sharing (DMS) Policy, which applies to all new and ongoing NIH-funded research in the IRP, as of January 25, 2023, that is associated with a ZIA, with a clinical protocol that undergoes scientific review and/or will involve genomic data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available as soon as possible or at the time of associated publication. Data not published in a manuscript will be shared via public source once the data set completes QC.
Access Criteria: Clinical data will be made available upon request and with the permission of the study PI. Genomic data are made available via dbGAP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_002363-C.html